CLINICAL TRIAL: NCT04411264
Title: Evaluation of the Effect of Virtual Reality on Pain in the Management of Chronic Wounds: Multicentric Randomized Controlled Trial.
Brief Title: Evaluation of the Effect of Virtual Reality on Pain in the Management of Chronic Wounds.
Acronym: DouReV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/CHU/12
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Chronic Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic protocol for pain management (No Intervention): classic protocol for pain management during chronic wound dressing
- Virtual reality for pain management (Experimental): protocol associating virtual reality with the classic protocol for pain management during the treatment of chronic wound dressings
  Interventions: Device: virtual reality

INTERVENTIONS:
Device: virtual reality — Use of a virtual reality headset while caring for chronic wound dressings
  Arms: Virtual reality for pain management

SUMMARY:
Pain management is a priority axis of health insurance spending objectives and contributes to improving the quality of care.There are several types of pain: acute, chronic and induced. These are often found in the management of chronic wounds. The high prevalence of chronic wounds represents a major public health problem. Chronic wounds require long, painful and regular treatment. When dressing these wounds, pain management is essential. Indeed, it can generate healing delays. Usually, pharmacological methods are used to reduce the pain induced by care. But these methods can lead to undesirable effects. Thus, new non-pharmacological techniques are emerging.The investigators therefore wish to assess the effect of virtual reality on pain induced by care during the repair of dressings in the management of chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Knowing how to read and write French
* Able to understand the issues of the study and give consent
* Carrier of a chronic wound (ulcers, bedsores or wounds of the diabetic foot)
* Requiring a weekly dressing treatment in the department for at least 4 successive treatments(4 weeks)
* With pain during pre-inclusion care at least ≥3 to the Visual Analog Scale
* Person with cognitive and sensory capacities adapted to Virtual Reality (pre-inclusion verification on a device test of 5 to 10 minutes)
* Person affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Carriers of a wound located on the face or end of the head and interfering with the proper use of the Virtual Reality mask
* Visually impaired and / or hard of hearing impacting the correct use of the Virtual Reality mask (test of 5 to 10 minutes of the device during the pre-inclusion visit)
* Patient not fluent in French.
* Current diagnosis of epilepsy, dementia or other neurological diseases preventing the use of Virtual Reality hardware and software
* Patients under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-induced pain | 4 weeks
  (AVS) Analog Visual Scale 0 to 10 : 0 for no pain ; 10 for maximum pain imaginable

SECONDARY OUTCOMES:
Level of situational anxiety | 4 weeks
  (STAI-Y-A) State-Trait Anxiety Scale - Overall score varies between 20 and 80. The higher the score, the more anxious the patient.
Duration of treatment | 4 weeks
  time in seconds
Worse Treatment-induced pain | 4 weeks
  Analog Visual Scale
Frequency of use of analgesic | 4 weeks
  analgesic consumption
Time spent thinking about pain | 4 weeks
  (AVS) Analog Visual Scale 0 to 10 : 0 for no thought of pain ; 10 for throughout the treatment
Healing process | 4 weeks
  measurement of the wound on photograhies by imageJ ® planimetry software
Medical Outcome Study Short Form | 4 weeks
  (SF6) Short Form (36) Health Survey_ Quality of life questionnaire
Tolerance of virtual reality | 4 weeks
  frequency of occurrence and intensity of motion sickness events

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Centre Hospitalier Universitaire de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No